CLINICAL TRIAL: NCT01628107
Title: A Phase III, Open-label, Multicenter, Long-term Safety Study Of Intravenous Epoetin Hospira In Patients With Chronic Renal Failure Requiring Hemodialysis And Receiving Epoetin Maintenance Treatment
Brief Title: A Phase 3, Long-Term Safety Study of Intravenous Epoetin Hospira in Patients With Chronic Renal Failure Requiring Hemodialysis and Receiving Epoetin Maintenance Treatment. AiME - Anemia Management With Epoetin
Acronym: AiME - 03
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPOE-11-03; C3461004 (Other: Alias Study Number)
Record Dates: First submitted 2012-06-22; First posted 2012-06-26 (Estimated); Results first posted 2018-07-19 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-06

CONDITIONS: Chronic Renal Failure Requiring Hemodialysis
Keywords: Chronic renal failure; hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Epoetin Hospira (Experimental): Epoetin Hospira will be administered by IV bolus injection 1 to 3 times per week per each patient's dosing schedule. Other ESAs (except for long-acting) may be used as rescue therapy.
  Interventions: Biological: Epoetin Hospira

INTERVENTIONS:
Biological: Epoetin Hospira — Intravenous (IV) injection
  Other Names: ESA; Erythropoetin Stimulating Agent

SUMMARY:
The purpose of the study is to determine the long-term safety in treatment-emergent adverse events (TEAEs) of intravenous (IV) administration of Epoetin Hospira for maintenance of target hemoglobin (Hgb) levels in patients treated for anemia associated with chronic renal failure and on hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is able to provide written Informed Consent after the risks and benefits of the study have been explained prior to any study-related activities.
2. Patient previously completed the core study Treatment Period up to and including Week 24 study assessments per protocol and is willing to continue open-label Epoetin Hospira for up to 48 weeks.
3. If female, patient must be postmenopausal for at least 1 year prior to enrollment, surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy), or practicing at least 1 of the following methods of birth control:

   * Hormonal contraceptives (oral, parenteral, or transdermal) for at least 3 months prior to enrollment
   * Intrauterine device
   * Double-barrier method (condoms, contraceptive sponge, diaphragm, or vaginal ring with spermicidal jellies or cream)

   If hormonal contraceptives are used, the specific contraceptive must have been used for at least 3 months prior to enrollment. If the patient is currently using a hormonal contraceptive, she should also use a barrier method during this study and for at least 30 days following the administration of the patient's last open-label dose.
4. Adequate methods of contraception to prevent pregnancy are to be maintained throughout the course of the study in both male and female study subjects.

Exclusion Criteria:

1. Patient had a serious or severe adverse event in the core study that, in the opinion of the Investigator, was probably or definitely related to epoetin use and precluded safe use of epoetin.
2. Any of the following that developed during the core study and prior to enrollment:

   * Myocardial infarction
   * Stroke (cerebrovascular accident)/cerebrovascular insult (minor stroke) or transient ischemic attack/intracerebral bleeding/cerebral infarction
   * Severe/unstable angina
   * Coronary angioplasty, bypass surgery, or peripheral artery bypass graft
   * Decompensated congestive heart failure (New York Heart Association [NYHA] class IV)
   * Pulmonary embolism
   * Deep vein thrombosis or other thromboembolic event
   * Received live or attenuated vaccination (except flu vaccination)
3. A patient with any active, uncontrolled systemic, inflammatory, or malignant disease that developed during the core study and in the Investigator's opinion may be significant to exclude participation in the study, including but not limited to demyelinating diseases such as multiple sclerosis, microbial, viral, or fungal infection or mental disease.
4. Any newly developed significant drug sensitivity or a significant allergic reaction to any drug, as well as known hypersensitivity or idiosyncratic reaction to epoetin (or its excipients, including albumin) or any other related drugs that in the judgment of the Investigator is exclusionary for study participation.
5. A female patient who is pregnant, lactating, or planning a pregnancy during the study.
6. History of drug abuse or alcohol abuse during the core study prior to enrollment as determined by the Investigator.
7. Current participation or participation in a drug or other investigational research study within 30 days prior to enrollment (except the core study or any observational studies with prior written approval from Hospira).
8. May not be able to comply with the requirements of this clinical study, communicate effectively with study personnel, or is considered by the Investigator, for any reason, to be an unsuitable candidate for the study.
9. Evidence of human immunodeficiency virus (HIV) or hepatitis B surface antigen (HBsAg).
10. A patient who, in the Investigator's opinion, has any clinically significant abnormal laboratory results that may impact patient safety.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2012-07-16 (Actual); Primary Completion 2015-01-02 (Actual); Study Completion 2015-01-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (110):
- United States (108):
  - North America Research Institute, Azusa, California
  - Bellflower Dialysis Center, Bellflower, California
  - National Institute of Clinical Research, Commerce, California
  - DaVita Premier Dialysis Center, Cudahy, California
  - Davita - South Valley Dialysis, Encino, California
  - Ong, Rubin, Shahmir A Medical Corp DBA: Solano Kidney Care, Fairfield, California
  - Fairfield Dialysis Center, Fairfield, California
  - Renal Consultants Medical Group, Granada Hills, California
  - Advanced Medical Research (Administrative), Lakewood, California
  - Long Beach Clinical Trials, Long Beach, California
  - Westcoast Dialysis, Long Beach, California
  - DaVita Bixby Knolls Dialysis, Long Beach, California
  - United Dialysis Center, Long Beach, California
  - Long Beach Dialysis, Long Beach, California
  - Imperial Care Dialysis Center, Lynwood, California
  - Kidney Research Center, Lynwood, California
  - Modesto Kidney Center, Modesto, California
  - Novo Research d/b/a Foundation Research, Modesto, California
  - Parkway Kindey Center, Modesto, California
  - Oakdale Kidney Center, Oakdale, California
  - National Institute of Clinical Research, Ontario, California
  - Ontario Dialysis Center, Ontario, California
  - Paramount Dialysis Center, Paramount, California
  - Sierra View Dialysis Center, Porterville, California
  - Sierra View District Hospital Dialysis Center, Porterville, California
  - Sierra View District Hospital, Porterville, California
  - Sierra View Nephrology, Inc., Porterville, California
  - Nephrology Educational Services and Research, Inc, Tarzana, California
  - Santa Clarita Kidney Center, Valencia, California
  - American Institute of Research, Whittier, California
  - Santa Fe Springs Dialysis, Whittier, California
  - Nephrology and Hypertension Associates,PC, Middlebury, Connecticut
  - Waterbury Dialysis Center, Waterbury, Connecticut
  - Greater Waterbury Dialysis, Waterbury, Connecticut
  - Innovative Medical Research of South Florida, Inc,, Aventura, Florida
  - West Boca Dialysis Center, Boca Raton, Florida
  - Florida Kidney Center, Lauderhill, Florida
  - South Florida Research Institute, Laureda Lake, Florida
  - Coconut Creek Dialysis JV, Margate, Florida
  - American Renal Associates Naples Dialysis Center, Naples, Florida
  - Innovative Medical Research of South Florida, Inc., North Miami Beach, Florida
  - Physicians Dialysis of North Beach, North Miami Beach, Florida
  - Discovery Medical Research Group, Inc.,, Ocala, Florida
  - Discovery Medical Research Group, Inc., Ocala, Florida
  - Ocala Regional Kidney Center, East, Ocala, Florida
  - Silver Springs Shores Dialysis Center, Ocala, Florida
  - Ft. Lauderdale Kidney Center, Plantation, Florida
  - Plantation Kidney Center, Plantation, Florida
  - Tamarac Kidney Center, Tamarac, Florida
  - Dialysis of Dublin, Dublin, Georgia
  - Renal Physicians of Georgia, PC, Dublin, Georgia
  - Liberty Dialysis/Boise Kidney & Hypertension Institute, Caldwell, Idaho
  - Liberty Dialysis/Boise Kidney & Hypertension Institute, Meridian, Idaho
  - Pacific Renal Research Institute/Boise Kidney & Hypertension Institute, Meridian, Idaho
  - Liberty Dialysis/Boise Kidney & Hypertension Institute, Nampa, Idaho
  - Neomedica South, Chicago, Illinois
  - FMC Ross Englewood Dialysis, Chicago, Illinois
  - Neomedica Evergreen Park, Evergreen Park, Illinois
  - Research by Design, LLC, Evergreen Park, Illinois
  - North Suburban Nephrology, LLC, Gurnee, Illinois
  - Neomedica Round Lake, Round Lake, Illinois
  - Clinton Township Dialysis, Clinton Township, Michigan
  - Grosse Pointe Dialysis, Detroit, Michigan
  - Renaissance Renal Research Institute, LLC, Detroit, Michigan
  - Biloxi Dialysis, Biloxi, Mississippi
  - FMC/South Mississippi Kidney Center of Gulfport, Gulfport, Mississippi
  - South Mississippi Medical Research, PLLC, Gulfport, Mississippi
  - Barnes-Jewish Dialysis Center, St Louis, Missouri
  - Chromalloy American Kidney Center Washington University School of Medicine, St Louis, Missouri
  - Lower Manhattan Dialysis Center II, New York, New York
  - Mountain Kidney and Hypertension Associates, P A, Asheville, North Carolina
  - Asheville Kidney Center, Asheville, North Carolina
  - ECU Nephrology and Hypertension, Greenville, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Cincinnati VA Medical Center, Cincinnati, Ohio
  - Fresenius Greater Columbus Regional Dialysis Center, Columbus, Ohio
  - HNC Dialysis, Ltd., Columbus, Ohio
  - Delaware Valley Nephrology and Hypertension Associates, PC, Philadelphia, Pennsylvania
  - Fresenius Medical Care- Mt. Airy Kidney Center, Philadelphia, Pennsylvania
  - Fresenius Medical Care - Olney Dialysis Center, Philadelphia, Pennsylvania
  - Anderson Dialysis Clinic, Anderson, South Carolina
  - AnMed Health, Anderson, South Carolina
  - Nephrology and Internal Medicine of Anderson, Anderson, South Carolina
  - Columbia Nephrology Associates, P. A., Columbia, South Carolina
  - Columbia Nephrology Associates, PA, Columbia, South Carolina
  - Fresenius Medical Care Columbia JV, Columbia, South Carolina
  - Fresenius Medical Care Meadowlake JV, Columbia, South Carolina
  - Fresenius Medical Care South Columbia JV, Columbia, South Carolina
  - Fresenius Medical Care SE Columbia JV, Columbia, South Carolina
  - Sumter Dialysis Clinic, Sumter, South Carolina
  - Gamma Medical Research Inc., Edinburg, Texas
  - Med Center Dialysis, Houston, Texas
  - Fresenius Medical Care Kidney Center, Houston, Texas
  - Meyerland Dialysis, Houston, Texas
  - Millennium Clinical Research, Inc., Houston, Texas
  - Southwest Houston Dialysis, Houston, Texas
  - DaVita North Park, Houston, Texas
  - North Shepherd Dialysis Center, Houston, Texas
  - Southwest Houston Research, Ltd., Houston, Texas
  - Dialysis Center of Lubbock, Lubbock, Texas
  - Fresenius Medical Care McAllen, McAllen, Texas
  - Fresenius Medial Care Mission, Mission, Texas
  - Missouri City Dialysis, Missouri City, Texas
  - NW Medical Center DaVita Dialysis, San Antonio, Texas
  - San Antonio Kidney Disease Center Physicians Group, P.L.L.C., San Antonio, Texas
  - Floyd Curl DaVita Dialysis Center, San Antonio, Texas
  - Butler Farm Dialysis, Hampton, Virginia
  - Peninsula Kidney Associates, Hampton, Virginia
- Puerto Rico (2):
  - Consolidated Medical Plaza, Caguas
  - Fresenius Medical Care·Humacao, Humacao

REFERENCES:
- [Derived] Wish JB, Rocha MG, Martin NE, Reyes CRD, Fishbane S, Smith MT, Nassar G. Long-term Safety of Epoetin Alfa-epbx for the Treatment of Anemia in ESKD: Pooled Analyses of Randomized and Open-label Studies. Kidney Med. 2019 Aug 28;1(5):271-280. doi: 10.1016/j.xkme.2019.06.009. eCollection 2019 Sep-Oct. PMID 32734207

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with chronic renal failure were receiving Epoetin maintenance therapy in study EPOE-10-01 (NCT01473407) prior to enrollment and treatment in the current study.
Groups:
- Epoetin Hospira: Participants were enrolled to receive Epoetin Hospira intravenous injection 1 to 3 times every week over a period of 48 weeks. Dose was adjusted to maintain the hemoglobin (Hb) level from 9 to 11 gram per deciliter (g/dL).
Period: Overall Study
Arm/Group | Epoetin Hospira
Started | 414
Treated | 406
Completed | 295
Not Completed | 119
Not completed — Withdrawal by Subject | 17
Not completed — Lost to Follow-up | 4
Not completed — Adverse Event | 33
Not completed — Physician Decision | 2
Not completed — Not met Inclusion/Exclusion Criteria | 1
Not completed — Non-compliant with Study Procedures | 10
Not completed — Not Treated | 8
Not completed — Sponsor Decision | 11
Not completed — Missed Study Drug More than 2 Weeks | 7
Not completed — Relocated | 8
Not completed — Kidney Transplant | 9
Not completed — Use of Standard of Care | 9

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Arm/Group | Epoetin Hospira
Number analyzed (Participants) | 406
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.45 (12.062)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 169
  Male | 237

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (AEs): Week 1
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment emergent are events that emerged during the treatment period and were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Up through 7 days after first dose of study drug (Week 1)
Population: Safety analysis set included all participants who received at least 1 dose of study drug. Here, "number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Epoetin Hospira
Number analyzed (Participants) | 400
Percentage of participants | 13.0

2. Primary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (AEs): Over Week 1 to 12
Description: as for outcome 1
Time Frame: Week 1 up to Week 12
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Epoetin Hospira
Number analyzed (Participants) | 406
Percentage of participants | 59.4

3. Primary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (AEs): Over Week 13 to 24
Description: as for outcome 1
Time Frame: Week 13 up to Week 24
Population: Safety analysis set included all participants who received at least 1 dose of study drug. Here, ''number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Epoetin Hospira
Number analyzed (Participants) | 369
Percentage of participants | 57.5

4. Primary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (AEs): Over Week 25 to 36
Description: as for outcome 1
Time Frame: Week 25 up to Week 36
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Epoetin Hospira
Number analyzed (Participants) | 339
Percentage of participants | 54.3

5. Primary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (AEs): Over Week 37 to 48
Description: as for outcome 1
Time Frame: Week 37 up to Week 48
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Epoetin Hospira
Number analyzed (Participants) | 315
Percentage of participants | 51.7

6. Primary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (AEs): Over Week 1 to 48
Description: as for outcome 1
Time Frame: Week 1 up to Week 48
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Epoetin Hospira
Number analyzed (Participants) | 406
Percentage of participants | 85.7

7. Secondary Outcome: Mean Weekly Dosage of Epoetin Hospira : Over Week 1 to 48
Time Frame: Week 1 up to Week 48
Population: Full analysis set (FAS) included all enrolled participants and had at least 1 dose of Epoetin Hospira study drug and had at least 1 Hb value. Here, "number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Unit per kilogram per week (U/kg/week)
Arm/Group | Epoetin Hospira
Number analyzed (Participants) | 400
Unit per kilogram per week (U/kg/week) | 95.30 (85.515)

8. Secondary Outcome: Mean Weekly Dosage of Epoetin Hospira for Interval of 12 Weeks
Time Frame: Week 1 up to Week 12; Week 13 up to Week 24; Week 25 up to Week 36; Week 37 up to Week 48
Population: FAS included all enrolled participants and had at least 1 dose of Epoetin Hospira study drug and had at least 1 Hb value.
Measure: Mean (Standard Deviation); unit: U/kg/week
Arm/Group | Epoetin Hospira
Number analyzed (Participants) | 403
U/kg/week
  Week 1 to Week 12: number analyzed (Participants) | 393
  Week 1 to Week 12 | 94.93 (89.219)
  Week 13 to Week 24: number analyzed (Participants) | 352
  Week 13 to Week 24 | 94.84 (89.303)
  Week 25 to Week 36: number analyzed (Participants) | 321
  Week 25 to Week 36 | 94.01 (86.0)
  Week 37 to Week 48: number analyzed (Participants) | 303
  Week 37 to Week 48 | 99.55 (95.510)

9. Secondary Outcome: Mean Hemoglobin Levels: Over Week 1 to 48
Time Frame: Week 1 up to Week 48
Population: FAS included all enrolled participants and had at least 1 dose of Epoetin Hospira study drug and had at least 1 Hb value. Here, "number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Epoetin Hospira
Number analyzed (Participants) | 402
g/dL | 10.21 (0.629)

10. Secondary Outcome: Mean Hemoglobin Levels for Interval of 12 Weeks
Time Frame: Week 1 up to Week 12; Week 13 up to Week 24; Week 25 up to Week 36; Week 37 up to Week 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Epoetin Hospira
Number analyzed (Participants) | 402
g/dL
  Week 1 to Week 12 | 10.26 (0.789)
  Week 13 to Week 24: number analyzed (Participants) | 364
  Week 13 to Week 24 | 10.25 (0.762)
  Week 25 to Week 36: number analyzed (Participants) | 339
  Week 25 to Week 36 | 10.18 (0.865)
  Week 37 to Week 48: number analyzed (Participants) | 314
  Week 37 to Week 48 | 10.21 (0.818)

11. Secondary Outcome: Mean Hematocrit Levels: Over Week 1 to 48
Description: Hematocrit is defined as the percentage of red blood cells in the blood.
Time Frame: Week 1 up to Week 48
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells
Arm/Group | Epoetin Hospira
Number analyzed (Participants) | 402
Percentage of red blood cells | 32.17 (2.164)

12. Secondary Outcome: Mean Hematocrit Levels for Interval of 12 Weeks
Description: Hematocrit is defined as the percentage of red blood cells in the blood.
Time Frame: Week 1 up to Week 12; Week 13 up to Week 24; Week 25 up to Week 36; Week 37 up to Week 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells
Arm/Group | Epoetin Hospira
Number analyzed (Participants) | 403
Percentage of red blood cells
  Week 1 to Week 12: number analyzed (Participants) | 402
  Week 1 to Week 12 | 32.26 (2.695)
  Week 13 to Week 24: number analyzed (Participants) | 364
  Week 13 to Week 24 | 32.21 (2.569)
  Week 25 to Week 36: number analyzed (Participants) | 339
  Week 25 to Week 36 | 32.03 (2.978)
  Week 37 to Week 48: number analyzed (Participants) | 314
  Week 37 to Week 48 | 32.17 (2.738)

13. Secondary Outcome: Percentage of Participants With Hemoglobin Level Outside the Target Range
Description: Percentage of participants with hemoglobin level outside the target range of 9.0 to 11.0 g/dL were reported.
Time Frame: Week 1 up to Week 48
Population: as for outcome 8
Measure: Number; unit: Percentage of participants
Arm/Group | Epoetin Hospira
Number analyzed (Participants) | 403
Percentage of participants | 90.1

14. Secondary Outcome: Percentage of Participants Who Received Blood Transfusions
Time Frame: Week 1 up to Week 48
Population: as for outcome 8
Measure: Number; unit: Percentage of participants
Arm/Group | Epoetin Hospira
Number analyzed (Participants) | 403
Percentage of participants | 9.7

15. Other Pre Specified Outcome: Percentage of Participants With Hemoglobin Level Less Than (<) 8.0 Gram Per Deciliter (g/dL)
Time Frame: Week 1 up to Week 48
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Epoetin Hospira
Number analyzed (Participants) | 402
Percentage of participants | 13.9

16. Other Pre Specified Outcome: Percentage of Participants With Hemoglobin Level Greater Than (>) 12.0 Gram Per Deciliter (g/dL)
Time Frame: Week 1 up to Week 48
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Epoetin Hospira
Number analyzed (Participants) | 402
Percentage of participants | 20.9

17. Other Pre Specified Outcome: Number of Participants With Clinically Significant Change From Baseline in Hemoglobin Levels
Description: Participants with clinically significant change from baseline in hemoglobin levels were upon investigator's discretion.
Time Frame: Baseline up to Week 48
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Epoetin Hospira
Number analyzed (Participants) | 406
Participants | 0

18. Other Pre Specified Outcome: Number of Participants Who Received Concomitant Medication
Time Frame: Week 1 up to Week 48
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Epoetin Hospira
Number analyzed (Participants) | 406
Participants | 406

19. Other Pre Specified Outcome: Number of Participants With Clinically Significant Change From Baseline in Laboratory Tests
Description: Laboratory tests included: Hematology (hematocrit, hemoglobin, red blood cells count, reticulocytes, white blood cells count, neutrophils, bands, lymphocytes, monocytes, basophils, eosinophils, platelets, mean corpuscular volume); Coagulation panel (prothrombin time, international normalized ratio, activated partial thromboplastin time); Chemistry (blood urine nitrogen, creatinine, total bilirubin, alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, sodium, potassium, magnesium, calcium, gamma-glutyl transpeptidase, phosphorus, uric acid, total protein, glucose, albumin, C-reactive protein); iron status (plasma ferritin, transferrin saturation). Participants with clinically significant change from baseline in laboratory tests were based on investigator's discretion.
Time Frame: Baseline up to Week 48
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Epoetin Hospira
Number analyzed (Participants) | 406
Participants | 0

20. Other Pre Specified Outcome: Number of Participants With Clinically Significant Change From Baseline in 12-Lead Electrocardiogram (ECG)
Description: ECG parameters included: PR interval, QRS complex, QT interval and QTC interval. Participants with clinically significant change from baseline in 12-lead ECGs were based on investigator's discretion.
Time Frame: Baseline up to Week 48
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Epoetin Hospira
Number analyzed (Participants) | 406
Participants | 2

21. Other Pre Specified Outcome: Number of Participants With Clinically Significant Change From Baseline in Physical Examinations
Description: Physical examination included examination of the skin, eyes, ears, nose, throat, head, neck, thyroid, lungs, chest, abdomen, extremities, lymphatic, cardiovascular, musculoskeletal and neurological systems. Participants for any clinically significant changes in physical examination were based on the investigator's discretion.
Time Frame: Baseline up to Week 48
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Epoetin Hospira
Number analyzed (Participants) | 406
Participants | 0

22. Other Pre Specified Outcome: Percentage of Participants With Anti-Recombinant Human Erythropoietin (Anti-rhEPO) Antibodies
Description: Percentage of participants with at least 1 positive anti-rhEPO antibody were reported. Radioimmunoprecipitation assay was used to determine the presence of anti-rhEPO antibodies.
Time Frame: Baseline, Week 48
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Epoetin Hospira
Number analyzed (Participants) | 406
Percentage of participants
  Baseline | 0
  Week 48: number analyzed (Participants) | 321
  Week 48 | 0.6

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study. Safety Population.
Arm/Group | Epoetin Hospira
Serious Adverse Events (participants affected / at risk) | 168/406
Other Adverse Events (participants affected / at risk) | 277/406
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Epoetin Hospira (N=406)
Anaemia (Blood and lymphatic system disorders) | 4
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Acute coronary syndrome (Cardiac disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 13
Angina pectoris (Cardiac disorders) | 7
Aortic valve incompetence (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 3
Bradycardia (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 6
Cardiac failure (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 10
Cardio-respiratory arrest (Cardiac disorders) | 7
Cardiomegaly (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 4
Coronary artery occlusion (Cardiac disorders) | 2
Hypertrophic cardiomyopathy (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 4
Myocardial ischaemia (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Ventricular fibrillation (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Gastrointestinal angiodysplasia (Congenital, familial and genetic disorders) | 1
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 1
Thyroid mass (Endocrine disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 2
Colitis (Gastrointestinal disorders) | 1
Colitis ischaemic (Gastrointestinal disorders) | 1
Colonic polyp (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 3
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3
Hiatus hernia (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 2
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 2
Small intestinal obstruction (Gastrointestinal disorders) | 2
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 3
Chest pain (General disorders) | 1
Death (General disorders) | 1
Non-cardiac chest pain (General disorders) | 3
Pyrexia (General disorders) | 1
Systemic inflammatory response syndrome (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 2
Cholecystitis acute (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 5
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Cellulitis (Infections and infestations) | 4
Osteomyelitis (Infections and infestations) | 4
Pneumonia (Infections and infestations) | 16
Sepsis (Infections and infestations) | 18
Staphylococcal sepsis (Infections and infestations) | 4
Abdominal abscess (Infections and infestations) | 1
Abscess limb (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 2
Appendicitis perforated (Infections and infestations) | 2
Arteriovenous fistula site infection (Infections and infestations) | 1
Arteriovenous graft site infection (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 3
Bronchitis (Infections and infestations) | 1
Cardiac valve abscess (Infections and infestations) | 1
Cellulitis staphylococcal (Infections and infestations) | 1
Cystitis escherichia (Infections and infestations) | 1
Device related infection (Infections and infestations) | 2
Device related sepsis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 3
Endocarditis (Infections and infestations) | 3
Gangrene (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 1
Infected skin ulcer (Infections and infestations) | 1
Influenza (Infections and infestations) | 2
Liver abscess (Infections and infestations) | 1
Lobar pneumonia (Infections and infestations) | 2
Localised infection (Infections and infestations) | 1
Mastoiditis (Infections and infestations) | 1
Staphylococcal bacteraemia (Infections and infestations) | 2
Nocardiosis (Infections and infestations) | 1
Otitis externa (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Peridiverticular abscess (Infections and infestations) | 1
Perirectal abscess (Infections and infestations) | 1
Pneumonia viral (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Sepsis syndrome (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Streptococcal bacteraemia (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 4
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 3
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 3
Clavicle fracture (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 4
Femur fracture (Injury, poisoning and procedural complications) | 2
Fibula fracture (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Splenic rupture (Injury, poisoning and procedural complications) | 1
Sternal fracture (Injury, poisoning and procedural complications) | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 1
Vascular graft complication (Injury, poisoning and procedural complications) | 1
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1
Vascular pseudoaneurysm ruptured (Injury, poisoning and procedural complications) | 1
Liver function test abnormal (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Diabetic foot (Metabolism and nutrition disorders) | 2
Fluid overload (Metabolism and nutrition disorders) | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 13
Hypoglycaemia (Metabolism and nutrition disorders) | 6
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Osteolysis (Musculoskeletal and connective tissue disorders) | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1
Breast cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-small cell lung cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 3
Metabolic encephalopathy (Nervous system disorders) | 3
Carotid artery stenosis (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Cerebral ischaemia (Nervous system disorders) | 1
Diabetic hyperosmolar coma (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Haemorrhage intracranial (Nervous system disorders) | 1
Hemiparesis (Nervous system disorders) | 1
Hepatic encephalopathy (Nervous system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 2
Mental impairment (Nervous system disorders) | 2
Presyncope (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 3
Transient ischaemic attack (Nervous system disorders) | 1
Unresponsive to stimuli (Nervous system disorders) | 2
Delirium (Psychiatric disorders) | 1
Hallucination (Psychiatric disorders) | 1
Azotaemia (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 2
Renal failure chronic (Renal and urinary disorders) | 1
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1/169 — This event was gender specific event.
Vaginal haemorrhage (Reproductive system and breast disorders) | 1/169 — This event was gender specific event.
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
Accelerated hypertension (Vascular disorders) | 1
Aortic stenosis (Vascular disorders) | 1
Arterial thrombosis limb (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hypertension (Vascular disorders) | 6
Hypertensive crisis (Vascular disorders) | 3
Hypertensive emergency (Vascular disorders) | 2
Hypotension (Vascular disorders) | 2
Haematoma (Vascular disorders) | 1
Ischaemic limb pain (Vascular disorders) | 1
Malignant hypertension (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1
Peripheral ischaemia (Vascular disorders) | 1
Peripheral vascular disorder (Vascular disorders) | 1
Vascular occlusion (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Epoetin Hospira (N=406)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 81
Nausea (Gastrointestinal disorders) | 58
Headache (Nervous system disorders) | 51
Diarrhoea (Gastrointestinal disorders) | 49
Dizziness (Nervous system disorders) | 47
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 42
Hypotension (Vascular disorders) | 41
Vomiting (Gastrointestinal disorders) | 39
Cough (Respiratory, thoracic and mediastinal disorders) | 36
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 35
Pyrexia (General disorders) | 35
Oedema peripheral (General disorders) | 33
Anaemia (Blood and lymphatic system disorders) | 25
Pain in extremity (Musculoskeletal and connective tissue disorders) | 24
Hypertension (Vascular disorders) | 22
Asthenia (General disorders) | 21
Back pain (Musculoskeletal and connective tissue disorders) | 21
Constipation (Gastrointestinal disorders) | 21
Upper respiratory tract infection (Infections and infestations) | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single centre publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.